CLINICAL TRIAL: NCT06275113
Title: BRING-UP Prevention
Status: Recruiting | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K25
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Heart Disease; Cerebrovascular Disorders; Peripheral Arterial Disease
MeSH Terms: conditions — Myocardial Ischemia; Cerebrovascular Disorders; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to assess in patients with a documented athero-thrombotic event: coronary artery disease (CAD), cerebrovascular disease (CVD), peripheral artery disease (PAD):

* the level of adherence to guideline recommendations with the assumption to improve the rate of patients at goal for cholesterol levels.
* the level of adherence to guideline recommendations and the rate of patients at goal for the other relevant and modifiable risk factors for cardiovascular event recurrence.

DETAILED DESCRIPTION:
Observational, prospective, multicenter study conducted in a large, representative sample of Italian cardiology centers.

Phases:

1. First educational intervention to discuss the recommendations of guidelines for secondary prevention strategies.
2. Data collection for 3 months or up to 30 consecutive patients in patients with documented CAD/CVD/PAD on a web Case Record Form (CRF) generating warning on the most relevant guideline recommendations, and, when guidelines are not followed, asking the reason for non-adherence.
3. Evaluation of the primary and secondary end-points of the study at 6 months after enrollment.
4. Second educational intervention to share the results of the first enrollment period of the study focusing the attention on existing gaps between guidelines recommendations and clinical practice.
5. New data collection for 3 months or up to 30 consecutive patients in patients with documented CAD/CVD/PAD on a web CRF generating warning on the most relevant guideline recommendations, and, when guidelines are not followed, asking the reason for non-adherence.
6. Additional evaluation of the primary and secondary end-points of the study at 6 months after enrollment.
7. 12-month follow-up for all patients included in both enrolment phases.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes at birth, age ≥18 years

At least one of the following clinical conditions:

* Documented CAD defined as:

  * Prior Acute Coronary Syndrom (ACS)
  * Prior Coronary Artery Bypass Graft (CABG)
  * Prior Percutaneous Coronary Intervention (PCI)
* Documented PAD (previous peripheral bypass surgery or angioplasty, limb or foot amputation, intermittent claudication with objective evidence of peripheral artery disease, Ankle Brachial Index (ABI)<90).
* Documented CVD: Ischemic stroke, previous carotid vascular interventions.
* Signed informed consent.

Exclusion Criteria:

* Active neoplasia or very severe disease compromising short-medium term life expectancy.
* Participation in interventional studies.
* Patients already enrolled into the study from another participating center or in the previous enrolling phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients discharged (after ordinary hospitalisation or day hospital) or managed as outpatients with a documented prior athero-thrombotic event: coronary artery disease (CAD), cerebrovascular disease (CVD), peripheral artery disease (PAD).
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to guideline for cholesterol level | 6 months
  Rate of patients at goal for LDL cholesterol (<55 mg/dL)

SECONDARY OUTCOMES:
Adherence to guideline for other risk factors | 6 months
  Rate of patients at goal for BP (SBP/DBP < 130/80 mmHg) and at goal for HbA1c (<7%) as well as rate of overweight patients (BMI > 27 kg/m2) who show a weight loss of at least 10%

OTHER OUTCOMES:
Patients' outcome | 12 months
  Rate of occurrence of clinical events (all-cause deaths, recurrent athero-thrombotic events, all cause hospitalizations, specific causes of death and hospitalizations) during the 12 follow-up of each enrolment phase.

CONTACTS AND LOCATIONS:
Locations (196):
- Italy (196):
  - Ospedale Barone Lombardo - Cardiologia E Utic, Canicattì, AG
  - Ospedale San Giacomo D'Altopasso - Uoc Cardiologia, Licata, AG
  - Ospedale Santo Spirito - Sc Cardiologia, Casale Monferrato, AL
  - Ospedale San Giacomo - Sc Cardiologia, Novi Ligure, AL
  - Ospedali Riuniti - Clinica Di Cardiologia E Aritmologia, Ancona, AN
  - Ospedali Riuniti - Sod Cardiologia Ospedaliera E Utic, Ancona, AN
  - Casa Di Cura Villa Serena - U.O. Cardiologia Riabilitativa, Iesi, AN
  - Ospedale Madonna Del Soccorso - Uoc Cardiologia Indirizzo Riabilitativo, San Benedetto del Tronto, AP
  - Ospedale San Donato - U.O.C Cardiologia, Arezzo, AR
  - Ospedale Valdichiana Santa Margherita - Uosd Cardiologia S.O. Cortona, Cortona, AR
  - Aorn San Giuseppe Moscati - U.O. Cardiologia/Utic 'D. Rotiroti', Avellino, AV
  - Ospedale Miulli - U.O.C. Cardiologia - Utic, Acquaviva delle Fonti, BA
  - Ospedale Della Murgia - Fabio Perinei - S.C. Cardiologia-Utic, Altamura, BA
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Ics Maugeri Spa Societa' Benefit Irccs Bari - Cardiologia Riabilitativa, Bari, BA
  - Mater Dei Hospital - Riabilitazione Cardiologica, Bari, BA
  - Ospedale Umberto I - U.O.C. Cardiologia, Corato, BA
  - Ospedale San Giacomo - Uoc Cardiologia, Monopoli, BA
  - Ospedale Degli Infermi - Sc Di Cardiologia, Ponderano, BI
  - Presidio Ospedaliero "Santa Maria Del Prato" - U.O.C. Di Cardiologia-Utic, Feltre, BL
  - Ospedale Di Bentivoglio - U.O. Cardiologia Pianura, Bentivoglio, BO
  - Ospedale Maggiore - U.O.C. Di Cardiologia, Bologna, BO
  - Ospedale Bellaria - U.O. Di Cardiologia, Bologna, BO
  - Ospedale Perrino - U.O.C. Di Cardiologia, Brindisi, BR
  - Casa Di Cura San Camillo - U.O. Cardiologia, Brescia, BS
  - Ospedale Di Desenzano Del Garda - Divisione Di Cardiologia - U.C.C., Desenzano del Garda, BS
  - Ospedale Civile 'La Memoria' - U.O. Di Cardiologia, Gavardo, BS
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Lumezzane - U.O. Di Cardiologia Riabilitativa, Lumezzane, BS
  - Ospedale Monsignor Angelo R. Di Miccoli - Uoc Cardiologia/Utic, Barletta, BT
  - Ospedale Centrale Bolzano - Cardiologia E Prove Funzionali, Bolzano, BZ
  - Arnas G. Brotzu - Cardiologia Con Utic, Cagliari, CA
  - Arnas G. Brotzu - S.S.D. Cardioriabilitazione, Cagliari, CA
  - A.O.U. Cagliari Policlinico Monserrato - Sc Cardiologia Utic Emodinamica, Monserrato, CA
  - Azienda Ospedaliera S. Anna E S. Sebastiano - U.O. Cardiologia D'Emergenza Con Utic, Caserta, CE
  - Villa Delle Magnolie - Riabilitazione Cardiologica, Castel Morrone, CE
  - Casa Di Cura San Michele - Uo Cardiologia, Maddaloni, CE
  - Ospedale San Giuseppe E Melorio - U.O.C. Cardiologia Utic, Santa Maria Capua Vetere, CE
  - Ospedale Policlinico Ss. Annunziata - Uoc Cardiologia-Utic, Chieti, CH
  - Santa Barbara Hospital - Cardiologia, Gela, CL
  - Azienda Ospedaliera Santa Croce E Carle - Sc Cardiologia, Cuneo, CN
  - Ospedale Regina Montis Regalis - U.O. Cardiologia-Utic, Mondovì, CN
  - Ospedale Maggiore Ss. Annunziata - Sc Cardiologia, Savigliano, CN
  - Ospedale Oglio Po - U.O. Di Cardiologia-Utic, Casalmaggiore, CR
  - Ospedale Annunziata - Uoc Cardiologia Interventistica, Cosenza, CS
  - Ospedale Spoke Paola- Cetraro Po Paola - Utic Cardiologia, Paola, CS
  - Policlinico Di Catania Presidio San Marco - Cardiologia Utic, Catania, CT
  - P.O. Garibaldi-Nesima - Arnas Garibaldi - U.O.C. Di Cardiologia Con Utic, Catania, CT
  - P.O. "Materdomini" - A.O.U. "Renato Dulbecco" - Ssd Cardiologia Riabilitativa, Catanzaro, CZ
  - Ospedale G.B. Morgagni - L. Pierantoni - U.O. Cardiologia, Forlì, FC
  - Arcispedale Sant'Anna - U.O. Cardiologia, Ferrara, FE
  - Policlinico Riuniti - S.C. Di Cardiologia Universitaria-Utic, Foggia, FG
  - San Francesco Hospital - U.O.C. Cardiologia, Foggia, FG
  - Ospedale Casa Sollievo Della Sofferenza - Cardiologia - Utic - Riabil Cardiologica, San Giovanni Rotondo, FG
  - Aou Careggi - Riabilitazione Cardiologica, Florence, FI
  - E.O. Ospedali Galliera - S. C. Cardiologia E U.T.I.C., Genova, GE
  - Ospedale San Giovanni Di Dio - Sc Cardiologia (Gorizia-Monfalcone), Gorizia, GO
  - Ospedale Civile San Polo - Sc Cardiologia (Gorizia-Monfalcone), Monfalcone, GO
  - Presidio Ospedaliero - U.O. Cardiologia, Sanremo, IM
  - Ospedale Alessandro Manzoni - S.C. Di Cardiologia, Lecco, LC
  - Presidio Ospedaliero F. Ferrari - Ssd Cardiologia - Utic, Casarano, LE
  - Ospedale San Giuseppe Da Copertino - U.O. Di Cardiologia, Copertino, LE
  - Ospedale Vito Fazzi - Uoc Cardiologia-Utic Ed Emodinamica, Lecce, LE
  - Ospedale Ignazio Veris Delli Ponti - Uoc Cardiologia-Utic "E. Vilei", Scorrano, LE
  - Ospedali Riuniti - U.O.C. Cardiologia E Utic, Livorno, LI
  - Istituto 'Marco Pasquali' Icot - Riabilitazione Cardiologica, Latina, LT
  - Nuovo Ospedale Versilia - Sc Cardiologia, Camaiore, LU
  - Ospedale Giovanni Paolo Ii - Uosd Utic, Policoro, Matera
  - Ospedale Pio Xi - U.O.C. Di Cardiologia, Desio, MB
  - Fondazione Irccs San Gerardo Dei Tintori - Ospedale San Gerardo - U.O.C. Cardiologia, Monza, MB
  - Ospedale Di Seregno - Riabilitazione Specialistica Cardiologica, Seregno, MB
  - Nuovo Ospedale Di Vimercate - S.C. Cardiologia E Utic, Vimercate, MB
  - Ospedale Generale Provinciale - U.O. Cardiologia, Macerata, MC
  - Iomi Istituto Ortopedico F. Scalabrino - Uo Cardiologia, Messina, ME
  - Irccs Centro Neurolesi Bonino Pulejo - P.O Piemonte - Cardiologia E Utic, Messina, ME
  - Azienda Ospedaliera Papardo - U.O. Cardiologia Con Utic - Emodinamica, Messina, ME
  - Ospedale Di Cernusco Sul Naviglio - U. O. Di Cardiologia E Ucc, Cernusco sul Naviglio, MI
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico - Uoc Malattie Cardiovascolari, Milan, MI
  - Centro Cardiologico Monzino Irccs - Terapia Intensiva Cardiologica (Utic), Milan, MI
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Milano - Riabilitazione Cardiologica, Milan, MI
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Milano - Uo Cure Subacute, Milan, MI
  - Irccs Santa Maria Nascente Fond. Don Gnocchi - Cardiologia Riabilitativa, Milan, MI
  - ASST SANTI PAOLO E CARLO - PO San Carlo - CARDIOLOGIA-UCC, Milan, MI
  - Irccs Ospedale Galeazzi - Sant'Ambrogio - Cardiologia Universitaria Ed Imaging Cardiaco, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Diagnosi E Cure Terr. Malattie Cardiache, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 1 - Emodinamica, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 4 - Diagnostica E Riabilitativa, Milan, MI
  - Presidio Ospedaliero Di Passirana - Cardiologia Riabilitativa, Rho, MI
  - Irccs Policlinico San Donato - Cardiologia Riabilitativa, San Donato Milanese, MI
  - Irccs Policlinico Multimedica - Uo Di Cardiologia, Sesto San Giovanni, MI
  - Ospedale Citta' Di Sesto San Giovanni - Sc Cardiologia-Ucc Asst Nord Milano (Bassini-Ssg), Sesto San Giovanni, MI
  - Ospedale Santa Maria Bianca - U.O. Di Cardiologia, Mirandola, MO
  - Ospedale Civile Di Baggiovara - U.O. Di Cardiologia, Modena, MO
  - Ospedale Di Sassuolo - Cardiologia, Sassuolo, MO
  - Ospedale San Giovanni Di Dio - Uo Cardiologia - Utic, Frattamaggiore, Napoli
  - Fondazione G. Giglio - U.O. Di Cardiologia, Cefalù, PA
  - Ospedale Buccheri La Ferla Fatebenefratelli - Ssd Riabilitazione Cardiovascolare, Palermo, PA
  - Aou Policlinico P. Giaccone - U.O.C. Cardiologia, Palermo, PA
  - Arnas P.O. Civico E Benfratelli - Uoc Utic, Palermo, PA
  - Maria Eleonora Hospital - Cardiologia, Palermo, PA
  - Aor Villa Sofia-Cervello P.O. Cervello - U.O. Cardiologia - Cervello, Palermo, PA
  - Aor Villa Sofia-Cervello Po Villa Sofia - Uoc Cardiologia E Utic E Emodinamica -Villa Sofia, Palermo, PA
  - Ospedale Unico Della Val Tidone - Cardiologia E Riabilitazione, Castel San Giovanni, PC
  - Ospedale Civile 'Guglielmo Da Saliceto' - Uoc Cardiologia E Utic, Piacenza, PC
  - Ospedale Di Cittadella - U.O. Cardiologia, Cittadella, PD
  - Ospedale Civile Dello Spirito Santo - Cardiologia Con Utic, Pescara, PE
  - Presidio Ospedaliero Citta' Di Castello - U.O. Cardiologia/Utic, Città di Castello, PG
  - Ospedale Gubbio-Gualdo Tadino - U.O. Di Utic E Cardiologia, Gubbio, PG
  - Azienda Ospedaliera Di Perugia - S.C. Cardiologia, Perugia, PG
  - Ospedale Ss. Cosma E Damiano - Sos Cardiologia, Pescia, Pistoia
  - Ospedale Ss. Cosma E Damiano - Sos Riabilitazione Cardiologica, Pescia, Pistoia
  - Ftgm - Stabilimento Di Pisa - Cardiologia E Medicina Cardiovascolare, Pisa, PI
  - Auxilium Vitae Volterra - Riabilitazione Cardiologica, Volterra, PI
  - Presidio Ospedaliero Per La Salute Di Sacile - Cardiologia Preventiva E Riabilitativa, Sacile, PN
  - Ospedale Di S. Vito Al Tagliamento - Ssd Cardiologia San Vito - Spilimbergo, San Vito al Tagliamento, PN
  - Ospedale Civile - U.O.C. Cardiologia - Utic, Fidenza, PR
  - Istituto Don Gnocchi - U.O. Prevenzione E Riabilitazione Cardiovascolare, Parma, PR
  - Presidio Ospedaliero San Salvatore - Cardiologia E Utic, Pesaro, PU
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Pavia - U.O. Di Riabilitazione Cardiologica, Pavia, PV
  - Ospedale Civile - U.O. Di Cardiologia, Voghera, PV
  - Ospedale Civile - Uo Servizio Cardiologia, Lugo, RA
  - Ospedale Civile Santa Maria Delle Croci - Uoc Cardiologia, Ravenna, RA
  - Ospedale Civile Di Guastalla - Sos Cardiologia E Riabilitazione Card Area Nord, Guastalla, RE
  - Ospedale E. Franchini - S.O.S. Cardiologia, Montecchio Emilia, RE
  - Po Santa Maria Nuova - Ausl Re Irccs - Soc Cardiologia Ospedaliera, Reggio Emilia, RE
  - Ospedale Riccardo Guzzardi - U.O.C. Di Cardiologia-Utic, Vittoria, RG
  - P.O. San Camillo de Lellis - U.O.C. Cardiologia, Rieti, RI
  - Ospedali Riuniti Anzio-Nettuno - U.O.C. Di Cardiologia - Utic, Anzio, RM
  - Ospedale Dei Castelli - U.O.C. Di Cardiologia E Utic, Ariccia, RM
  - Ospedale Civile San Paolo - U.O.C. Cardiologia - Utic, Civitavecchia, RM
  - Ospedale L. Parodi Delfino - U.O.C. Di Cardiologia - Utic, Colleferro, RM
  - Icr Villa Delle Querce - Riabilitazione Cardiorespiratoria, Nemi, RM
  - P.O. San Filippo Neri - Asl Roma 1 - Cardiologia Clinica E Riabilitativa, Roma, RM
  - Inmi Lazzaro Spallanzani Irccs - Servizio Di Cardiologia Del Dipartimento Clinico, Roma, RM
  - Ospedale San Camillo - Uoc Cardiologia, Roma, RM
  - Ospedale Sandro Pertini - Uoc Cardiologia, Roma, RM
  - Ospedale Sandro Pertini - Uosd Cardiologia D'Urgenza, Roma, RM
  - Fondazione Policlinico Universitario A. Gemelli Irccs - Uosd Cardiologia D'Urgenza, Roma, RM
  - Policlinico Casilino - U.O.C. Cardiologia, Roma, RM
  - Osp. Fatebenefratelli Isola Tiberina - Uoc Cardiologia Diagnostica Interventistica-Utic, Roma, RM
  - Ospedale Sant'Andrea Di Roma - U.O.C. Cardiologia, Roma, RM
  - Ospedale Santo Spirito - Uoc Cardiologia, Roma, RM
  - Ospedale San Giovanni Evangelista - U.O.C. Di Cardiologia - Utic, Tivoli, RM
  - Ospedale Infermi - U.O. Cardiologia, Rimini, RN
  - Ospedale Maria Ss. Addolorata - U.O. Di Cardiologia Utic, Eboli, SA
  - Presidio Ospedaliero Umberto I - Uoc Cardiologia - Utic, Nocera Inferiore, SA
  - Presidio Ospedaliero Luigi Curto - Uo Cardiologia-Utic, Polla, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Cardiologia Intensiva Ospedaliera, Salerno, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Ssd Utic, Salerno, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Uoc Clinica Cardiologica, Salerno, SA
  - Ospedale Villa Malta - Cardiologia E Utic, Sarno, SA
  - Ospedale San Luca - U.O. Utic - Cardiologia, Vallo della Lucania, SA
  - Aou Senese Ospedale S. Maria Alle Scotte - Cardiologia, Siena, SI
  - Ospedale San Bartolomeo - Sc Riabilitazione Cardiologica, Sarzana, SP
  - P.O. Lentini - Uosd Di Cardiologia Con Utic, Lentini, SR
  - Ospedale Ss. Annunziata - Cardiologia Clinica Ed Interventistica, Sassari, SS
  - Po Ponente - Ospedale Santa Corona - Sc Cardiologia Ponente, Pietra Ligure, SV
  - Casa Di Cura Villa Verde - Cardiologia, Taranto, TA
  - Osp. San Pancrazio-Santo Stefano - Riabilitazione Cardiologica, Arco, TN
  - Ospedale Santa Chiara - Divisione Di Cardiologia, Trento, TN
  - Por Cirie' Lanzo Presidio Cirie' - S.C. Cardiologia, Cirié, TO
  - Aou San Luigi Gonzaga - S.C.D.O. Cardiologia, Orbassano, TO
  - Casa Di Cura Villa Serena - Riabilitazione Cardiorespiratoria, Piossasco, TO
  - Ospedale Degli Infermi - Sc Cardiologia, Rivoli, TO
  - Ospedale San Giovanni Bosco - Sc Cardiologia, Torino, TO
  - Casa Di Cura Pineta Del Carso - U.O. Riabilitazione Cardiologica, Duino-Aurisina, TS
  - Asugi Trieste - Sc Patologie Cardiovascolari, Trieste, TS
  - Pou "Santa Maria Della Misericordia" - S.O.C. Cardiologia, Udine, UD
  - Ospedale Multimedica Castellanza - Cardiologia, Castellanza, VA
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale Di Circolo Galmarini - Cardiologia, Tradate, VA
  - Ospedale Sant'Andrea - Sc Cardiologia, Vercelli, VC
  - Ospedale Dell'Angelo - U.O.C. Cardiologia, Mestre, VE
  - Policlinico San Marco - Riabilitazione Cardiologica, Mestre, VE
  - Ospedale P.F. Calvi - Uos Di Cardiologia Riabilitativa, Noale, VE
  - Ospedale Civile - U.O.C. Di Cardiologia, San Donà di Piave, VE
  - Ospedale Civile - U.O.C. Di Cardiologia, Arzignano, VI
  - Ospedale Alto Vicentino - U.O.C. Cardiologia - Ucic, Santorso, VI
  - Ospedale Civile San Bortolo - U.O.C. Cardiologia, Vicenza, VI
  - Irccs Ospedale Sacro Cuore Don Calabria - U.O. Di Cardiologia, Negrar, VR
  - Ospedale G. Fracastoro - U.O.C. Di Cardiologia, San Bonifacio, VR
  - Aoui Di Verona - U.O. Cardiologia, Verona, VR
  - Ospedale Belcolle - Uoc Cardiologia Ed Emodinamica, Viterbo, VT
  - Ospedale Ss. Trinita' - S.C. Di Cardiologia, Borgomanero
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Veruno - Uo Cardiologia Riabilitativa, Gattico
  - Presidio Ospedaliero San Giugliano - U.O. Cardiologia - Utic, Giugliano in Campania
  - Ospedale Madonna Delle Grazie - Ssd Utic, Matera
  - Ospedale Buon Consiglio Fatebenefratelli - U.O.Complessa Di Cardiologia E Utic, Napoli
  - Aorn Cardarelli - U.O. Cardiologia Con Utic, Napoli
  - Aorn Ospedale Dei Colli - P.O. Monaldi - Uosd Malattie Cardiologiche Congenite Adulti-Guch, Napoli
  - Ospedale Dei Pellegrini - Uoc Cardiologia-Utic, Napoli
  - Ospedale S. Giovanni Bosco - Sc Cardiologia - Utic, Napoli
  - Ospedale Del Mare - U.O. Cardiologia Con Utic-Emodinamica, Napoli
  - Aou Maggiore Della Carita' - Scdo Cardiologia Ii, Novara
  - Clinica San Gaudenzio - Uoa Cardiologia, Novara
  - Ospedale Santa Maria Delle Grazie - U.O. Cardiologia - Utic Con Emodinamica, Pozzuoli
  - Ospedale Mauriziano Umberto I - Sc Cardiologia, Torino